CLINICAL TRIAL: NCT05497362
Title: A Randomized Controlled Trial Study of the Use of Transcranial Direct Current Stimulation (tDCS) in Treating Dysarthria Post-stroke
Brief Title: Non-invasive Brain Stimulation as a Treatment for Dysarthria Post-stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence M.W. Ng, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW16-126
Record Dates: First submitted 2022-07-23; First posted 2022-08-11 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Dysarthria; Stroke
MeSH Terms: conditions — Dysarthria; Stroke

STUDY DESIGN:
Intervention Model Description: Double-blinded
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real tDCS (Experimental): Group 1 (n = 5) received anodal tDCS stimulation and intensive speech and voice therapy; tDCS and speech therapy was applied in 10 daily sessions during a 2-week period, administered on Monday to Friday. The anodal stimulation was delivered to the primary motor cortex (SM1) of the orofacial area.
  Interventions: Device: Real tDCS
- Sham tDCS (Sham Comparator): Group 2 (n = 4) received sham tDCS stimulation and intensive speech and voice therapy. For the sham tDCS group, the same setting of tDCS electrodes was applied on the scalp, but the stimulation only lasted for 30 sec in order to cause a similar sensation on the scalp. tDCS and speech therapy was applied in 10 daily sessions during a 2-week period, administered on Monday to Friday.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Real tDCS — 2mA of tDCS was delivered to the orofacial area of the primary motor cortex (SM1) for 15 minutes. Speech therapy was delivered simultaneously.
  Arms: Real tDCS
Device: Sham tDCS — 2mA of tDCS was delivered to the orofacial area of the primary motor cortex (SM1) for 30 sec. Speech therapy was delivered simultaneously.
  Arms: Sham tDCS

SUMMARY:
The proposed study aimed to determine if tDCS can help post-stroke patients with dysarthria.

DETAILED DESCRIPTION:
A total of 9 Cantonese-speaking chronic post-stroke patients who are suffering from dysarthria was recruited and randomly divided into treatment group and sham group. For the treatment group, an anodal high-definition tDCS of 2 milliampere (mA) lasting for 15 minutes was delivered to the primary motor cortex (SM1) in 10 daily sessions during a 2-week period. For the sham tDCS group, the same setting of tDCS electrodes was applied on the scalp, but the stimulation only lasted for 30 sec in order to cause similar sensation on the scalp as the other group. Simultaneous to the tDCS stimulation, both groups will receive speech and voice therapy for 30 minutes.

An array of outcome measures reflecting speech production ability including acoustic, kinematic, perceptual and self-perceptual qualities was obtained before and after stimulation. It was anticipated that post-stroke dysarthric patients will see improvement in speech production after stimulation. The results provided important insights into the effects of tDCS on articulatory movement in individuals with dysarthria post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* Cantonese-speaking adults
* At least 6 months after their initial stroke
* Dysarthria post-stroke

Exclusion Criteria:

* A personal or family history of epilepsy or seizures
* A history of another neurological condition
* Speech disorders
* Voice disorders
* Oro-maxillo-facial surgery involving the tongue and/or lip
* Severe cognitive impairment
* Severe aphasia
* Heart disease
* Metallic foreign body implant
* On medications that lower neural thresholds (e.g. tricyclines, antidepressants, neuroleptic agents, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Perceptual speech assessments | Change before and after tDCS stimulation at immediately post-treatment
  All participants were required to produce a sustained vowel /a/, repeated some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/), produce some single words, read a standard paragraph in Cantonese and had a two-minute conversation with the investigator. A professional grade microphone (SM58, Shure, USA) was used to record the speech production. Experienced speech-language pathologists blinded to the neurological condition and history of each participant analyzed the speech samples independently using a perceptual rating scale including 21 speech dimensions covering eight categories, including pitch, loudness, voice quality, resonance, rate, articulation, tone, and general impression. The speech samples were rated using a seven-point equal-appearing interval scale, with a "1" indicating within typical limit performance and a "7" severely deviated from the normal.
Acoustic measurement: Fundamental frequency (F0) | Change before and after tDCS stimulation at immediately post-treatment
  Fundamental frequency (F0) was obtained from sustained vowel phonation.
Acoustic measurement: Frequency perturbation (jitter %) | Change before and after tDCS stimulation at immediately post-treatment
  Frequency perturbation (jitter %) was obtained from sustained vowel phonation.
Acoustic measurement: Intensity perturbation (shimmer %) | Change before and after tDCS stimulation at immediately post-treatment
  Intensity perturbation (shimmer %) was obtained from sustained vowel phonation.
Acoustic measurement: Noise to harmonic ratio (NHR) | Change before and after tDCS stimulation at immediately post-treatment
  Noise to harmonic ratio (NHR) was obtained from sustained vowel phonation.
Acoustic measurement: Harmonic to noise ratio (HNR) | Change before and after tDCS stimulation at immediately post-treatment
  Harmonic to noise ratio (HNR) was obtained from sustained vowel phonation.

SECONDARY OUTCOMES:
Kinematic measurement: Duration | Change before and after tDCS stimulation at immediately post-treatment
  The lip and tongue function during speech production were traced real time and objectively measured using an electromagnetic articulography. All participants were required to produce single-syllable real words of consonant-vowel (CV) construction at high level tone embedded in a carrier phrase and repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/). A custom-written analysis programme was used to annotate and calculate the kinematic measures, including duration (ms), distance (mm), maximum velocity (mm/s), maximum acceleration (m/s2) and maximum deceleration (m/s2) in the approach (movement towards the upper lip/palate) and release (movement away from the upper lip/palate) phases along the z-axis, i.e., along the mid-sagittal plane.
Kinematic measurement: Distance | Change before and after tDCS stimulation at immediately post-treatment
  The lip and tongue function during speech production were traced real time and objectively measured using an electromagnetic articulography. All participants were required to produce single-syllable real words of consonant-vowel (CV) construction at high level tone embedded in a carrier phrase and repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/). A custom-written analysis programme was used to annotate and calculate the kinematic measures, including duration (ms), distance (mm), maximum velocity (mm/s), maximum acceleration (m/s2) and maximum deceleration (m/s2) in the approach (movement towards the upper lip/palate) and release (movement away from the upper lip/palate) phases along the z-axis, i.e., along the mid-sagittal plane.
Kinematic measurement: Maximum velocity | Change before and after tDCS stimulation at immediately post-treatment
  The lip and tongue function during speech production were traced real time and objectively measured using an electromagnetic articulography. All participants were required to produce single-syllable real words of consonant-vowel (CV) construction at high level tone embedded in a carrier phrase and repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/). A custom-written analysis programme was used to annotate and calculate the kinematic measures, including duration (ms), distance (mm), maximum velocity (mm/s), maximum acceleration (m/s2) and maximum deceleration (m/s2) in the approach (movement towards the upper lip/palate) and release (movement away from the upper lip/palate) phases along the z-axis, i.e., along the mid-sagittal plane.
Kinematic measurement: Maximum acceleration | Change before and after tDCS stimulation at immediately post-treatment
  The lip and tongue function during speech production were traced real time and objectively measured using an electromagnetic articulography. All participants were required to produce single-syllable real words of consonant-vowel (CV) construction at high level tone embedded in a carrier phrase and repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/). A custom-written analysis programme was used to annotate and calculate the kinematic measures, including duration (ms), distance (mm), maximum velocity (mm/s), maximum acceleration (m/s2) and maximum deceleration (m/s2) in the approach (movement towards the upper lip/palate) and release (movement away from the upper lip/palate) phases along the z-axis, i.e., along the mid-sagittal plane.
Kinematic measurement: Maximum deceleration | Change before and after tDCS stimulation at immediately post-treatment
  The lip and tongue function during speech production were traced real time and objectively measured using an electromagnetic articulography. All participants were required to produce single-syllable real words of consonant-vowel (CV) construction at high level tone embedded in a carrier phrase and repeat some syllables (i.e., /pa/, /ta/, /ka/ and /pataka/). A custom-written analysis programme was used to annotate and calculate the kinematic measures, including duration (ms), distance (mm), maximum velocity (mm/s), maximum acceleration (m/s2) and maximum deceleration (m/s2) in the approach (movement towards the upper lip/palate) and release (movement away from the upper lip/palate) phases along the z-axis, i.e., along the mid-sagittal plane.

CONTACTS AND LOCATIONS:
Overall Officials: Manwa L Ng, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No